CLINICAL TRIAL: NCT01858701
Title: Visual Performance Investigation of Two Toric Soft Contact Lenses
Acronym: CARDINAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A01335; P/438/13/L
Record Dates: First submitted 2013-05-17; First posted 2013-05-21 (Estimated); Results first posted 2014-10-22 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: Refractive Error; Astigmatism; Myopia; Hyperopia
Keywords: myopia; hyperopia; astigmatism; contact lenses
MeSH Terms: conditions — Refractive Errors; Astigmatism; Myopia; Hyperopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AO for Astig / Biofinity Toric (Other): Lotrafilcon B toric contact lenses worn in Period 1, followed by comfilcon A toric contact lenses in Period 2, as randomized. Each product will be worn bilaterally on a daily wear basis for 30 days, removed nightly. A minimum 1-day washout of no contact lens wear will precede each wear period.
  Interventions: Device: Lotrafilcon B toric contact lens; Device: Comfilcon A toric contact lens
- Biofinity Toric / AO for Astig (Other): Comfilcon A toric contact lenses worn in Period 1, followed by lotrafilcon B toric contact lenses in Period 2, as randomized. Each product will be worn bilaterally on a daily wear basis for 30 days, removed nightly. A minimum 1-day washout of no contact lens wear will precede each wear period.
  Interventions: Device: Lotrafilcon B toric contact lens; Device: Comfilcon A toric contact lens

INTERVENTIONS:
Device: Lotrafilcon B toric contact lens — Commercially available, silicone hydrogel contact lens for correction of astigmatism
  Other Names: AIR OPTIX® for ASTIGMATISM
Device: Comfilcon A toric contact lens — Commercially available, silicone hydrogel contact lens for correction of astigmatism
  Other Names: Biofinity® Toric

SUMMARY:
The purpose of this study is to compare the amount of coma as measured by aberrometry induced by two silicone hydrogel toric lenses in astigmatic participants.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent;
* Wears toric soft contact lenses;
* Can be successfully fit with study lenses within the power ranges available;
* Has cylinder of ≥ -0.75 diopter in both eyes;
* Has correctable vision of at least 0.1 (logMAR) or better in each eye at distance with both study lenses;
* Willing and able to wear study lenses on a daily wear basis for at least 5 days a week, minimum 8 hours per day, and attend all study visits;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any ocular condition that would contraindicate contact lens wear;
* Use of medications for which contact lens wear could be contraindicated;
* Monocular (only 1 eye with functional vision) or fit with 1 lens;
* History of herpetic keratitis, ocular surgery, or irregular cornea;
* Known sensitivity to the diagnostic pharmaceuticals to be used in the study;
* Requires presbyopic correction;
* Use of rewetting/lubricating eye-drops more than twice a day;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2013-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessie Lemp, MS, Study Director — Alcon Research; Lyndon Jones, PhD, Principal Investigator — School of Optometry and Vision Science

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 1 study center located in Canada.
Pre-assignment Details: Of the 49 enrolled, 9 participants were exited as screen failures prior to randomization. This reporting group includes all randomized participants (40).
Groups:
- AO for Astig / Biofinity Toric: Lotrafilcon B toric contact lenses worn in Period 1, followed by comfilcon A toric contact lenses in Period 2.
- Biofinity Toric / AO for Astig: Comfilcon A toric contact lenses worn in Period 1, followed by lotrafilcon B toric contact lenses in Period 2.
Period: Period 1, First 30 Days of Wear
Arm/Group | AO for Astig / Biofinity Toric | Biofinity Toric / AO for Astig
Started | 20 | 20
Completed | 20 | 19
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout Period, 1-13 Days
Arm/Group | AO for Astig / Biofinity Toric | Biofinity Toric / AO for Astig
Started | 20 | 19
Completed | 18 | 17
Not Completed | 2 | 2
Not completed — Inclusion/Exclusion Criteria Not Met | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2
Period: Period 2, Second 30 Days of Wear
Arm/Group | AO for Astig / Biofinity Toric | Biofinity Toric / AO for Astig
Started | 18 | 17
Completed | 18 | 16
Not Completed | 0 | 1
Not completed — Comfort | 0 | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all enrolled participants.
Groups:
- Overall: Lotrafilcon B toric contact lenses and comfilcon A toric contact lenses worn during Period 1 and Period 2 in a crossover assignment.
Arm/Group | Overall
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Mean Ocular Coma Score at 5mm Pupil at Day 30
Description: Ocular coma is a type of optical aberration or a distortion in image formation occurring when a bundle of light rays enters an optical system (eye) that is not parallel to the optic axis. Ocular coma will be measured in micrometers using a Ladarwave aberrometer. A lower number indicates less coma/less image distortion. One eye (right eye) contributed to the mean.
Time Frame: Day 30
Population: This analysis population includes all participants who completed the study.
Measure: Mean (Standard Deviation); unit: micrometers
Groups:
- Air Optix for Astig: Lotrafilcon B toric contact lenses worn bilaterally on a daily wear basis (removed nightly) during Period 1 or Period 2, for 30 days.
- Biofinity Toric: Comfilcon A toric contact lenses worn bilaterally on a daily wear basis (removed nightly) during Period 1 or Period 2, for 30 days.
Arm/Group | Air Optix for Astig | Biofinity Toric
Number analyzed (Participants) | 34 | 34
micrometers | 0.16 (0.09) | 0.24 (0.11)

ADVERSE EVENTS:
Time Frame: Adverse Events (AE) were collected for the duration of the study (5 months). An AE was defined as any undesirable medical occurrence which occurs in an individual participating in a clinical trial, whether or not it is considered to be trial-related.
Description: This analysis population includes all participants dispensed with study products, based on treatment-specific exposure.
Arm/Group | Air Optix for Astig | Biofinity Toric
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/38
Other Adverse Events (participants affected / at risk) | 0/37 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.